CLINICAL TRIAL: NCT03371966
Title: The Effects of Chronic Dietary Nitrate Supplementation on Constant Work Rate Exercise in High Functioning Middle Aged and Older Adults
Brief Title: Nitrate and Exercise Performance in Middle to Older Aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Isagenix International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WFU-IRB00022914
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Aging
Keywords: Beetroot Juice; Older Adults; Nitrate; Nitrite; Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Nitrate Beetroot Juice (Active Comparator): Beetroot juice high in nitrate will contain approximately 10.0 mmole nitrate per 120 ml.
  Interventions: Dietary Supplement: High Nitrate Beetroot Juice
- Low Nitrate Beetroot Juice (Placebo Comparator): Beetroot juice low in nitrate will contain approximately 0.5 mmole nitrate per 120 ml.
  Interventions: Dietary Supplement: Low Nitrate Beetroot Juice

INTERVENTIONS:
Dietary Supplement: High Nitrate Beetroot Juice — High nitrate beetroot juice (120 ml) will be administered for 7 days consecutively followed by a 7 day washout period then 7 consecutive days of low nitrate beetroot juice.
  Arms: High Nitrate Beetroot Juice
Dietary Supplement: Low Nitrate Beetroot Juice — Low nitrate beetroot juice (120 ml) will be administered for 7 days consecutively followed by a 7 day washout period then 7 consecutive days of high nitrate beetroot juice..
  Arms: Low Nitrate Beetroot Juice

SUMMARY:
Research with young healthy individuals has shown that beetroot juice beverages that contain large amounts of nitrate can improve exercise performance. Currently, it is not know whether the consumption of beetroot juice beverages high in nitrate can improve exercise performance in higher functioning middle- to older-aged adults. Therefore, the purpose of this study is to compare the effect of two different beetroot juice beverages (one high in nitrate and one low in nitrate) on exercise performance in middle- to older-aged adults.

DETAILED DESCRIPTION:
Nitric oxide (NO) has been identified as an important biological messenger involved in a number of physiological processes and is produced from L-arginine and molecular oxygen by NO-synthases or the more recently identified nitrate to nitrite to NO pathway. Dietary nitrate can be found in green leafy vegetables and is particularly abundant in beetroot and has been shown to be a potential ergogenic agent. The nitrate to nitrite to NO pathway has been shown to be involved in a number of physiological processes that could account for the improved exercise response following nitrate ingestion. However, the benefits of nitrate as an ergogenic aid have been shown to be effected by numerous factors that can influence its efficacy. These include age, training level, dosage and the mode, duration and intensity of the exercise.

Research with healthy younger moderately trained adults has repeatedly shown that ingestion of dietary nitrate can reduce the oxygen cost of submaximal exercise and improve exercise performance during high intensity exercise; whereas research with younger more highly trained endurance athletes is equivocal, since some studies have failed to demonstrate an improvement in exercise performance following nitrate ingestion.

The effects of nitrate have also been shown to be influenced by age. It has been documented that there are alterations in NO metabolism in older adults thought to result from impairment of the NO-synthases pathway. The investigators have shown that consumption of a supplement high in nitrate, such as beetroot juice, leads to elevated plasma nitrite levels and may help restore NO metabolism in older adults; whereas a diet high in nitrate without supplementation was insufficient at increasing plasma nitrite levels. The investigators research, along with that of others has shown nitrate supplementation to have positive effects in older adults with chronic diseases. However, research examining the effects of dietary nitrate on exercise performance in healthy older adults is scarce. Presently, it is unclear as to whether nitrate supplementation is beneficial to exercise performance in older adults and there is no data examining the effect of nitrate supplementation on exercise performance in active older adults. Therefore, the purpose of this study is to examine the effect of chronic nitrate supplementation on exercise performance in active higher functioning older adults.

ELIGIBILITY:
Inclusion Criteria:

* Competitive runner or cyclist.
* Able to pedal a stationary bike.
* Engage in moderate physical activity for at least 150 minutes per week or engage in strenuous physical activity for at least 75 minutes per week.
* Able to provide own transportation to study testing visits.
* Able to provide own transportation to study testing visits.
* Able to consume study beverages.
* Willingness to provide informed consent and participate in the intervention.

Exclusion Criteria:

* tobacco user (smoke or chew)
* participating in another intervention research study
* diabetes (type 1 or 2)
* atrophic gastritis
* hypo-or hyperthyroidism
* gout
* history of kidney stones
* history of hypotension
* aversion to the study-related testing procedures
* allergy/sensitivity/aversion to beetroot beverages
* medical conditions with contraindications for engaging in the vigorous aerobic exercise
* current treatment for cancer
* thyroid disorders,
* cardiovascular disease,
* chronic obstructive pulmonary disease,
* inflammatory bowel diseases
* impaired liver or kidney function
* taking phosphodiesterase type 5 inhibitors
* taking nitroglycerin or nitrate preparations
* taking proton pump inhibitors
* taking medication for hypothyroidism

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Constant Work Rate (CWR) Exercise Time | Seven days of treatment
  Exercise duration measured as the length of the exercise period at a submaximal exercise work rate.

SECONDARY OUTCOMES:
Isotime Oxygen Consumption (VO2) | Seven days of treatment
  VO2 during the constant work rate exercise test measured at the minimum exercise time from any of the tests (isotime).
Isotime Borg Rating of Perceived Exertion (RPE) | Seven days of treatment
  RPE during the constant work rate exercise test measured at the minimum exercise time from any of the tests (isotime).
Isotime Systolic Blood Pressure (Systolic BP) | Seven days of treatment
  Systolic BP during the constant work rate exercise test measured at the minimum exercise time from any of the tests (isotime).
Isotime Diastolic Blood Pressure (Systolic BP) | Seven days of treatment
  Diastolic BP during the constant work rate exercise test measured at the minimum exercise time from any of the tests (isotime).

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Berry, Ph.D., Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Gladwin MT. Role of the red blood cell in nitric oxide homeostasis and hypoxic vasodilation. Adv Exp Med Biol. 2006;588:189-205. doi: 10.1007/978-0-387-34817-9_17. PMID 17089890
- [Background] van Faassen EE, Bahrami S, Feelisch M, Hogg N, Kelm M, Kim-Shapiro DB, Kozlov AV, Li H, Lundberg JO, Mason R, Nohl H, Rassaf T, Samouilov A, Slama-Schwok A, Shiva S, Vanin AF, Weitzberg E, Zweier J, Gladwin MT. Nitrite as regulator of hypoxic signaling in mammalian physiology. Med Res Rev. 2009 Sep;29(5):683-741. doi: 10.1002/med.20151. PMID 19219851
- [Background] Jones AM. Dietary nitrate supplementation and exercise performance. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S35-45. doi: 10.1007/s40279-014-0149-y. PMID 24791915
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Background] Lansley KE, Winyard PG, Bailey SJ, Vanhatalo A, Wilkerson DP, Blackwell JR, Gilchrist M, Benjamin N, Jones AM. Acute dietary nitrate supplementation improves cycling time trial performance. Med Sci Sports Exerc. 2011 Jun;43(6):1125-31. doi: 10.1249/MSS.0b013e31821597b4. PMID 21471821
- [Background] Cermak NM, Gibala MJ, van Loon LJ. Nitrate supplementation's improvement of 10-km time-trial performance in trained cyclists. Int J Sport Nutr Exerc Metab. 2012 Feb;22(1):64-71. doi: 10.1123/ijsnem.22.1.64. PMID 22248502
- [Background] Miller GD, Marsh AP, Dove RW, Beavers D, Presley T, Helms C, Bechtold E, King SB, Kim-Shapiro D. Plasma nitrate and nitrite are increased by a high-nitrate supplement but not by high-nitrate foods in older adults. Nutr Res. 2012 Mar;32(3):160-8. doi: 10.1016/j.nutres.2012.02.002. PMID 22464802
- [Background] Berry MJ, Justus NW, Hauser JI, Case AH, Helms CC, Basu S, Rogers Z, Lewis MT, Miller GD. Dietary nitrate supplementation improves exercise performance and decreases blood pressure in COPD patients. Nitric Oxide. 2015 Aug 1;48:22-30. doi: 10.1016/j.niox.2014.10.007. Epub 2014 Oct 27. PMID 25445634
- [Background] Eggebeen J, Kim-Shapiro DB, Haykowsky M, Morgan TM, Basu S, Brubaker P, Rejeski J, Kitzman DW. One Week of Daily Dosing With Beetroot Juice Improves Submaximal Endurance and Blood Pressure in Older Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):428-37. doi: 10.1016/j.jchf.2015.12.013. Epub 2016 Feb 10. PMID 26874390
- [Derived] Berry MJ, Miller GD, Kim-Shapiro DB, Fletcher MS, Jones CG, Gauthier ZD, Collins SL, Basu S, Heinrich TM. A randomized controlled trial of nitrate supplementation in well-trained middle and older-aged adults. PLoS One. 2020 Jun 23;15(6):e0235047. doi: 10.1371/journal.pone.0235047. eCollection 2020. PMID 32574223